CLINICAL TRIAL: NCT00109811
Title: A Phase 2 Study of Prostate Specific Antigen Peptide 3A (PSA: 154-163(155L) ) (NSC # 722932, IND#9787) With Montanide ISA-51(NSC #675756, IND #9787) or Montanide® ISA 51 VG (NSC 737063) Vaccination in Prostate Cancer Recurrent
Brief Title: Vaccine Therapy in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02652; GCC-0430; CDR0000428259 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — prostate-specific antigen (154-163); Protein Subunit Vaccines; incomplete Freund's adjuvant; montanide ISA 51

ARMS (1):
- Treatment (Experimental): Patients receive PSA peptide vaccine (PSA-3A; PSA: 154-163 [155L]) emulsified in Montanide ISA-51 subcutaneously once in weeks 0, 2, 4, 6, 10, 14, and 18 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: PSA:154-163(155L) peptide vaccine; Biological: incomplete Freund's adjuvant; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: PSA:154-163(155L) peptide vaccine — Given subcutaneously
  Other Names: PSA PEP VAC; PSA-3A
Biological: incomplete Freund's adjuvant — Given subcutaneously
  Other Names: IFA; ISA-51; Montanide ISA 51
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well vaccine therapy works in treating patients with recurrent prostate cancer. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the T-lymphocyte immune response in patients with recurrent adenocarcinoma of the prostate treated with prostate-specific antigen (PSA) peptide vaccine (PSA-3A; PSA: 154-163 [155L]) emulsified in Montanide ISA-51.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this vaccine in these patients. II. Determine the effect of this vaccine on serum PSA level in these patients.

OUTLINE: This is a pilot study.

Patients receive prostate-specific antigen (PSA) peptide vaccine (PSA-3A; PSA: 154-163 [155L]) emulsified in Montanide ISA-51 subcutaneously once in weeks 0, 2, 4, 6, 10, 14, and 18 in the absence of disease progression* or unacceptable toxicity.

NOTE: *A rise in PSA alone is not considered disease progression.

After completion of study treatment, patients are followed at 1 and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Must have undergone radical prostatectomy ≥ 3 months ago
* Prostate-specific antigen (PSA) level ≥ 0.6 ng/mL and rising (after radical prostatectomy) on ≥ 2 measurements separated by ≥ 3 months
* HLA-A2-positive peripheral blood mononuclear cells by flow cytometry
* No clinical evidence of local recurrence

  * No palpable induration or mass in prostatic fossa
* No metastatic prostate cancer

  * No osseous metastases by bone scan
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* More than 1 year
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* Hepatitis B and C negative
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study PSA peptide vaccine or Montanide ISA-51
* No history of systemic autoimmune disease or autoimmune disease requiring anti-inflammatory or immunosuppressive therapy

  * Patients with history of autoimmune thyroiditis are eligible provided the patient requires only thyroid hormone replacement therapy AND disease has been stable for ≥ 1 year
* No known HIV positivity
* No ongoing or active infection
* No primary or secondary immune deficiency
* No psychiatric illness or social situation that would preclude study compliance
* No history of other uncontrolled illness
* No prior chemotherapy
* No prior hormonal therapy
* No concurrent systemic or ocular steroid therapy, except for any of the following:

  * Inhaled steroids for asthma
  * Limited topical steroids
  * Replacement doses of cortisone
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to the prostate

  * Prior radiotherapy to the pelvis after radical prostatectomy allowed
* See Disease Characteristics
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in frequency of CD8 T-lymphocyte precursors in peripheral blood mononuclear cells (PBMC), measured by ELISPOT assays | From baseline to 1 week after the last dose of study treatment
  A response is defined as at least a 5 fold higher frequency of INF-gamma secreting CD8 T cells after vaccination than before. A patient also will be considered a responder if no specific PSA: 154-163(155L) response was found before vaccination and a specific PSA: 154-163(155L) response is identified after vaccination.

SECONDARY OUTCOMES:
Effect of treatment on serum prostate-specific antigen level | Up to 4 weeks after completion of study treatment
  The PSA reduction is defined as is at least 50% fall in the serum PSA level after vaccination. The proportion of patients who showed a reduction in serum PSA will be estimated and corresponding 95% confidence intervals will be calculated.
Incidence of adverse events graded according to NCI CTCAE version 3.0 | Up to 4 weeks after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Alexander, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kouiavskaia DV, Berard CA, Datena E, Hussain A, Dawson N, Klyushnenkova EN, Alexander RB. Vaccination with agonist peptide PSA: 154-163 (155L) derived from prostate specific antigen induced CD8 T-cell response to the native peptide PSA: 154-163 but failed to induce the reactivity against tumor targets expressing PSA: a phase 2 study in patients with recurrent prostate cancer. J Immunother. 2009 Jul-Aug;32(6):655-66. doi: 10.1097/CJI.0b013e3181a80e0d. PMID 19483644